CLINICAL TRIAL: NCT00734968
Title: Does Prophylaxis With Macrobid Reduce the Incidence of Urinary Tract Infection in Patients Who Receive a Sub-Urethral Sling for the Treatment of Stress Urinary Incontinence: Randomized, Double Blinded Placebo Controlled Clinical Trial
Brief Title: Does Treatment With Macrobid Reduce Urinary Tract Infections in Patients Receiving a Sub-Urethral Sling for Incontinence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1108717
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Stress Incontinence
Keywords: Urinary tract infection (UTI); suburethral sling; Prevention; Nitrofurantoin; Prophylaxis
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Tract Infections | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Patients randomly assigned to be treated with nitrofurantoin 100mg PO BID x 3 days post-operatively
  Interventions: Drug: Nitrofurantoin
- Placebo (Placebo Comparator): Arm randomly assigned to receive placebo 1 tablet PO BID x 3 days post-operatively.The incidence of UTI in this group will be compared with group one (1)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitrofurantoin — Nitrofurantoin 100mg PO BID for 3 days post operatively following the placement of a sub-urethral sling for the treatment of stress urinary incontinence
  Other Names: Macrobid
  Arms: Treatment
Other: Placebo — 6 tablets to be taken 1 tablet PO BID. These tablets are identical to nitrofurantoin 100mg tablets.
  Arms: Placebo

SUMMARY:
This project will determine whether post-operative prophylaxis with macrobid will decrease the incidence of postoperative urinary tract infection in women receiving sub-urethral slings for the treatment of urinary incontinence.

DETAILED DESCRIPTION:
This project will be a randomized, double blinded, placebo controlled clinical trial. The aim of the trial is to determine whether or not post-operative prophylaxis with macrobid will decrease the incidence of postoperative urinary tract infection in women receiving sub-urethral slings for the treatment of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 who will undergo the placement of a sub-urethral sling for the treatment of stress urinary incontinence

Exclusion Criteria:

* Exclusion criteria are those with a known allergy to macrobid, those with glucose-6-phosphate deficiency, renal impairment, women breast feeding or with a known pregnancy, patients taking medications for gout, and those with known risk factors for complicated UTI (polycystic renal disease, nephrolithiasis, neurogenic bladder, diabetes, immuno-suppression, etc).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Jackson, M.D., Principal Investigator — University of Missouri-Columbia; Raymond T Foster, MD, MS, MHSc, Study Director — University of Missouri-Columbia
Locations (1):
- Scott and White Hosptial, Texas A&M University, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anger JT, Litwin MS, Wang Q, Pashos CL, Rodriguez LV. Complications of sling surgery among female Medicare beneficiaries. Obstet Gynecol. 2007 Mar;109(3):707-14. doi: 10.1097/01.AOG.0000255975.24668.f2. PMID 17329524
- [Background] Bent S, Nallamothu BK, Simel DL, Fihn SD, Saint S. Does this woman have an acute uncomplicated urinary tract infection? JAMA. 2002 May 22-29;287(20):2701-10. doi: 10.1001/jama.287.20.2701. PMID 12020306
- [Background] Aubin C. Evidence-based emergency medicine/rational clinical examination abstract. Does this woman have an acute uncomplicated urinary tract infection? Ann Emerg Med. 2007 Jan;49(1):106-8. doi: 10.1016/j.annemergmed.2006.09.022. No abstract available. PMID 17203544
- [Background] Bodelsson G, Henriksson L, Osser S, Stjernquist M. Short term complications of the tension free vaginal tape operation for stress urinary incontinence in women. BJOG. 2002 May;109(5):566-9. doi: 10.1111/j.1471-0528.2002.01195.x. PMID 12066948
- [Background] Ferro A, Byck D, Gallup D. Intraoperative and postoperative morbidity associated with cystoscopy performed in patients undergoing gynecologic surgery. Am J Obstet Gynecol. 2003 Aug;189(2):354-7; discussion 357. doi: 10.1067/s0002-9378(03)00677-x. PMID 14520192
- [Background] Grover ML, Bracamonte JD, Kanodia AK, Bryan MJ, Donahue SP, Warner AM, Edwards FD, Weaver AL. Assessing adherence to evidence-based guidelines for the diagnosis and management of uncomplicated urinary tract infection. Mayo Clin Proc. 2007 Feb;82(2):181-5. doi: 10.4065/82.2.181. PMID 17290725
- [Background] Gupta K, Hooton TM, Roberts PL, Stamm WE. Patient-initiated treatment of uncomplicated recurrent urinary tract infections in young women. Ann Intern Med. 2001 Jul 3;135(1):9-16. doi: 10.7326/0003-4819-135-1-200107030-00004. PMID 11434727
- [Background] Karram MM, Segal JL, Vassallo BJ, Kleeman SD. Complications and untoward effects of the tension-free vaginal tape procedure. Obstet Gynecol. 2003 May;101(5 Pt 1):929-32. doi: 10.1016/s0029-7844(03)00122-4. PMID 12738152
- [Background] Kuuva N, Nilsson CG. A nationwide analysis of complications associated with the tension-free vaginal tape (TVT) procedure. Acta Obstet Gynecol Scand. 2002 Jan;81(1):72-7. doi: 10.1034/j.1600-0412.2002.810113.x. PMID 11942891
- [Background] LaSala CA, Schimpf MO, Udoh E, O'Sullivan DM, Tulikangas P. Outcome of tension-free vaginal tape procedure when complicated by intraoperative cystotomy. Am J Obstet Gynecol. 2006 Dec;195(6):1857-61. doi: 10.1016/j.ajog.2006.06.060. PMID 17132487
- [Background] Lim JL, Quinlan DJ. Safety of a new transobturator suburethral synthetic sling (TVT-O) procedure during the training phase. J Obstet Gynaecol Can. 2006 Mar;28(3):214-217. doi: 10.1016/S1701-2163(16)32111-9. PMID 16650360
- [Background] Pugsley H, Barbrook C, Mayne CJ, Tincello DG. Morbidity of incontinence surgery in women over 70 years old: a retrospective cohort study. BJOG. 2005 Jun;112(6):786-90. doi: 10.1111/j.1471-0528.2004.00522.x. PMID 15924538
- [Background] Schraffordt Koops SE, Bisseling TM, Heintz AP, Vervest HA. Prospective analysis of complications of tension-free vaginal tape from The Netherlands Tension-free Vaginal Tape study. Am J Obstet Gynecol. 2005 Jul;193(1):45-52. doi: 10.1016/j.ajog.2004.11.004. PMID 16021057
- [Background] Sokol AI, Jelovsek JE, Walters MD, Paraiso MF, Barber MD. Incidence and predictors of prolonged urinary retention after TVT with and without concurrent prolapse surgery. Am J Obstet Gynecol. 2005 May;192(5):1537-43. doi: 10.1016/j.ajog.2004.10.623. PMID 15902154
- [Background] Tamussino KF, Hanzal E, Kolle D, Ralph G, Riss PA; Austrian Urogynecology Working Group. Tension-free vaginal tape operation: results of the Austrian registry. Obstet Gynecol. 2001 Nov;98(5 Pt 1):732-6. doi: 10.1016/s0029-7844(01)01565-4. PMID 11704161
- [Background] Tsivian A, Mogutin B, Kessler O, Korczak D, Levin S, Sidi AA. Tension-free vaginal tape procedure for the treatment of female stress urinary incontinence: long-term results. J Urol. 2004 Sep;172(3):998-1000. doi: 10.1097/01.ju.0000135072.27734.4a. PMID 15311022
- [Background] Valpas A, Kivela A, Penttinen J, Kauko M, Kujansuu E, Tomas E, Haarala M, Meltomaa S, Nilsson CK. Tension-free vaginal tape and laparoscopic mesh colposuspension in the treatment of stress urinary incontinence: immediate outcome and complications--a randomized clinical trial. Acta Obstet Gynecol Scand. 2003 Jul;82(7):665-71. PMID 12790850
- [Background] Ward K, Hilton P; United Kingdom and Ireland Tension-free Vaginal Tape Trial Group. Prospective multicentre randomised trial of tension-free vaginal tape and colposuspension as primary treatment for stress incontinence. BMJ. 2002 Jul 13;325(7355):67. doi: 10.1136/bmj.325.7355.67. PMID 12114234
- [Derived] Temtanakitpaisan T, Buppasiri P, Lumbiganon P, Laopaiboon M, Rattanakanokchai S. Prophylactic antibiotics for preventing infection after continence surgery in women with stress urinary incontinence. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD012457. doi: 10.1002/14651858.CD012457.pub2. PMID 35349162
- [Derived] Jackson D, Higgins E, Bracken J, Yandell PM, Shull B, Foster RT Sr. Antibiotic prophylaxis for urinary tract infection after midurethral sling: a randomized controlled trial. Female Pelvic Med Reconstr Surg. 2013 May-Jun;19(3):137-41. doi: 10.1097/SPV.0b013e318285ba53. PMID 23611930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 161 subjects were consecutively enrolled. 8 subjects were lost to protocol errors. 76 subjects were randomized to treatment and 77 to placebo. 1 subject from each arm was lost to follow up. 75 subjects in the treatment arm and 76 in the placebo arm were in the final analysis.
Groups:
- Placebo: Arm randomly assigned to receive placebo 1 tablet PO twice a day (BID) x 3 days post-operatively. The incidence of urinary tract infection (UTI) in this group will be compared with group one (1).
  Placebo: 6 tablets to be taken 1 tablet PO BID. These tablets are identical to nitrofurantoin 100 mg tablets.
Period: Overall Study
Arm/Group | Placebo | Treatment
Started | 77 | 76
Completed | 76 | 75
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 75 | 76 | 151
Age, Customized [Number; unit: participants]
  >18 years | 75 | 76 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 76 | 151
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 70 | 70 | 140
  Black | 1 | 1 | 2
  Hispanic | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 75 | 76 | 151

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-operative UTI Following the Placement of Sub-urethral Sling for the Treatment of Stress Urinary Incontinence
Description: The overall rate of UTI following the placement of sub-urethral sling for the treatment of stress urinary incontinence in our study was 24.8% (n = 37)
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 75 | 76
participants | 13 | 24

2. Primary Outcome: Incidence of Post-operative UTI in Placebo Group
Description: The incidence of UTI in the placebo group was 32%.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 75 | 76
participants | 13 | 24

3. Primary Outcome: Incidence of Post-operative UTI in Treatment Group
Description: The incidence of UTI in the nitrofurantoin group was 17.6%.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 75 | 76
participants | 13 | 24

ADVERSE EVENTS:
Arm/Group | Placebo | Treatment
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No